CLINICAL TRIAL: NCT02204917
Title: Contrast Enhanced Voiding Urosonography (ceVUS) With the Intravesical Administration of the Ultrasound Contrast Agent OPTISON TM (Trademark) for Vesicoureteral Reflux Detection and Urethral Imaging in Children.
Brief Title: CeVUS With Intravesical Administration of OPTISON TM (Trademark) in Children
Acronym: ceVUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kassa Darge (Other)
Responsible Party: Sponsor-Investigator, Kassa Darge, Sponsor-Investigator, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 13-010618
Record Dates: First submitted 2014-06-25; First posted 2014-07-31 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Vesico-Ureteral Reflux
Keywords: Ultrasound; Ultrasound Contrast Agents; Optison; contrast enhanced Voiding Urosonography (ceVUS); ceVUS; Vesicoureteral Reflux; Children; Kidney; Bladder; Urethra; Voiding Cystourethrography (VCUG); VCUG; Safety; Urinary tract
MeSH Terms: conditions — Vesico-Ureteral Reflux | interventions — FS 069

STUDY DESIGN:
Intervention Model Description: Comparative performance of contrast enhanced Voiding Urosonography (ceVUS) and Voiding Cystourethrography (VCUG) in the same participant and in the same session.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Comparative performance of ceVUS & VCUG (Experimental): Contrast enhanced Voiding Urosonography (ceVUS) will be performed with the intravesical administration of 0.1%-0.5% OPTISON / normal saline solution. The exact OPTISON dose (ml) that will be adjusted according to the age-related bladder filling capacity with a dose (ml) range from 0.3 mL in newborns to 3 mL in 18 year-old children. Voiding Cystourethrography (VCUG) exam will be subsequently performed using the same bladder catheter with intravesical administration of the x-ray contrast agent.
  Interventions: Drug: OPTISON

INTERVENTIONS:
Drug: OPTISON — Contrast enhanced Voiding Urosonography (ceVUS) with intravesical administration of OPTISON for vesicoureteral reflux detection and urethral imaging in children. Voiding Cystourethrography (VCUG) examination will be subsequently performed as part of the standard care.
  Other Names: Perflutren Protein-Type A Microspheres

SUMMARY:
In this clinical trial the investigators aim to evaluate the diagnostic feasibility and safety of ceVUS with the intravesical use of OPTISON for vesicoureteral reflux detection and urethral imaging in children.

DETAILED DESCRIPTION:
Contrast enhanced Voiding Urosonography (ceVUS) is a radiation free, highly sensitive imaging modality for vesicoureteral reflux (VUR) and urethral imaging in children. It employs ultrasound technology in combination with ultrasound contrast agent, which is administered intravesically via a bladder catheter. Currently, second generation ultrasound contrast agents are commercially available, comprising of gas-filled microbubbles. CeVUS in children is being widely practiced, primarily in Europe, despite the fact that none of the commercially available ultrasound contrast agents are yet approved for clinical applications in pediatric population. In the United States, there is limited clinical experience with ceVUS in children. Among the currently commercially available ultrasound contrast agents, OPTISON has already been used in research and off-label in clinical settings involving adults and children. One in-vitro study has been conducted aiming to optimize the ultrasound technical parameters and the dose of OPTISON for intravesical administration in children. In this clinical trial the investigators aim to evaluate the diagnostic feasibility and safety of ceVUS with the intravesical use of OPTISON for vesicoureteral reflux detection and urethral imaging in children.

ELIGIBILITY:
Inclusion criteria:

1. Children 2-18 years (first age cohort).
2. Children 0-18 years (second age cohort).
3. Referred to the Children's Hospital of Philadelphia (CHOP) for the performance of the clinically indicated Voiding Cystourethrography (VCUG) examination.
4. Parental/guardian permission (informed consent) and if appropriate, child's assent for additional performance of contrast enhanced Voiding Urosonography (ceVUS) examination.

Exclusion criteria:

1. Hypersensitivity to perflutren, blood, blood products or albumin.
2. Children requiring sedation for VCUG or ceVUS examinations.
3. Parents/guardians or subjects who, in the opinion of the principal investigator, may be non-compliant with study schedules or procedures.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kassa Darge, MD, PhD, Principal Investigator — Department of Radiology, the Children's Hospital of Philadelphia
Locations (1):
- Department of Radiology, the Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2014 to April 2015, the study team recruited and enrolled 31 eligible subjects scheduled for the clinically indicated voiding cysteourethrography (VCUG) examination from the daily inpatients/outpatients program of the Radiology Department at the Children's Hospital of Philadelphia.
Pre-assignment Details: One subject was enrolled into the study (informed consent signed), however, sedation was required as standard of care to perform the clinically indicated VCUG examination. Sedation constitutes an exclusion criterion. Therefore, this subject although enrolled into the study, did not actually complete it.
Groups:
- ceVUS With the Use of OPTISON & VCUG in the Same Session: OPTISON will be resuspended just before the performance of ceVUS examination, and 0.1%-0.5% of the bladder filling volume OPTISON / normal saline solution will be used for intravesical administration. The exact OPTISON dose (ml) will be adjusted according to the age-related bladder filling capacity with the maximum OPTISON dose (ml) range from 0.3 mL in newborns to 3 mL in 18 year-old children.
  VCUG exam will be performed using the same bladder catheter with intravesical administration of the x-ray contrast agent.
Period: Overall Study
Arm/Group | ceVUS With the Use of OPTISON & VCUG in the Same Session
Started | 31
Completed | 30
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- ceVUS With the Use of OPTISON & VCUG in the Same Session: OPTISON will be resuspended just before the performance of ceVUS examination, and 01%-0.5% OPTISON solution will be used for intravesical administration. The exact OPTISON dose (ml) will be adjusted according to the age-related bladder filling capacity with a maximum dose (ml) range from 0.3 mL in newborns to 3 mL in 18 year-old children. VCUG exam will be performed as part of the standard care using the same bladder catheter with intravesical administration of the x-ray contrast agent.
Arm/Group | ceVUS With the Use of OPTISON & VCUG in the Same Session
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Pelvic-ureter-units (PUUs) Detected With Vesicoureteral Reflux by Contrast Enhanced Voiding Urosonography (ceVUS) and by Voiding Cystourethrography (VCUG).
Description: 1. Presence or absence of vesicoureteral reflux identified by ceVUS and VCUG in each pelvic-ureter-unit (PUU) of each participant. PUU is an anatomic term that is used to describe the part of the urinary tract consisting of the renal calyces, pelvis and ureter.
  2. Grading the severity of reflux detected by ceVUS and VCUG. Grade 0: absence of reflux. If reflux is present, a 5 grade scale (grades I-V) is used to evaluate its severity. Grade I: reflux in the ureter, grade II: reflux up to the renal pelvis, grade III: reflux up to the renal pelvis with mild dilation of the ureter and pelvicalyceal system, grade IV reflux up to the renal pelvis with moderate dilation but preserved papillary impressions, grade V: reflux up to the renal pelvis with severe dilation and loss of papillary impressions. Higher grades of reflux are associated with increased risk of urinary tract infection.
  3. Imaging of the urethra during voiding (urethra visualized or not) and urethra pathology detection.
Time Frame: 10-15 minutes.
Population: In total, 59 kidneys with 62 pelvic-ureteric units (PUUs) in 30 children were analyzed.
Measure: Number; unit: pelvic-ureteric units (PUUs)
Units Other Than Participants: Number of Pelvic-Ureteric-Units (PUUs)
Groups:
- Severity of Reflux With ceVUS: Contrast enhanced Voiding Urosonography (ceVUS) OPTISON will be performed with the intravesical administration of 0.1%-0.5% OPTISON/normal saline solution. The exact OPTISON dose (ml) will be adjusted according to the age-related bladder filling capacity with a maximum dose (ml) range from 0.3 mL in newborns to 3 mL in 18 year-old children.
- Severity of Reflux With VCUG: Voiding Cystourethrography (VCUG) exam will be performed after ceVUS using the same bladder catheter with intravesical administration of the x-ray contrast agent.
Arm/Group | Severity of Reflux With ceVUS | Severity of Reflux With VCUG
Number analyzed (Participants) | 30 | 30
Number analyzed (Number of Pelvic-Ureteric-Units (PUUs)) | 62 | 62
pelvic-ureteric units (PUUs)
  Grade 0 reflux | 50 | 50
  Grade I reflux | 2 | 2
  Grade II reflux | 8 | 6
  Grade III reflux | 2 | 4
  Grade IV reflux | 0 | 0
  Grade V reflux | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events Following Contrast Enhanced Voiding Urosonography (ceVUS) With OPTISON and Voiding Cystourethrography (VCUG).
Description: The overall safety and tolerability of ceVUS with OPTISON was assessed before, during and immediately after each ceVUS and VCUG examinations, and in follow-up telephone interviews. Assessments included:
  1. evaluation of body systems for signs of generalized hypersensitivity, allergic or anaphylactoid reactions
  2. monitoring of heart rate and pulse oxygen saturation
  3. telephone questionnaire-based interview of parents/guardians and children 48 hours after the examinations for delayed adverse events.
  The severity of any possible adverse event was classified as mild, moderate or serious and the onset of symptoms was categorized as acute, subacute or delayed according to the World Health Organization (WHO) classifications. In addition, the adverse event was classified as anticipated if it was expected given the study related procedures or unanticipated if the subject was exposed to greater risk than previously known or recognized.
Time Frame: Within 1 hour and up to 2 days after ceVUS and VCUG examinations completion.
Measure: Number; unit: participants
Groups:
- ceVUS With the Use of OPTISON & VCUG in the Same Session: OPTISON will be resuspended just before the performance of ceVUS examination, 0.1%-0.5% OPTISON solution will be used for intravesical administration. The exact OPTISON dose (ml) will be adjusted according to the age-related bladder filling capacity with the maximum dose (ml) range from 0.3 mL in newborns to 3 mL in 18 year-old children. VCUG exam will be performed as part of the standard care using the same bladder catheter with intravesical administration of the x-ray contrast agent.
Arm/Group | ceVUS With the Use of OPTISON & VCUG in the Same Session
Number analyzed (Participants) | 30
participants
  Number of Participants without Adverse Events | 29
  Number of Participants with Adverse Events | 1

3. Secondary Outcome: Compare the Diagnostic Accuracy of Contrast Enhanced Voiding Urosonography (ceVUS) With Voiding CystoUrethroGraphy (VCUG) for Vesicoureteral Reflux Detection and Urethral Imaging in Children.
Description: The diagnostic accuracy of ceVUS will be assessed by evaluation of the true positive, true negative, false positive and false negative cases of reflux and urethral imaging findings detected by ceVUS and VCUG examinations.
Time Frame: 10-15 minutes.
Population: Voiding Cysteourethrography (VCUG) is used as the reference standard the results for ceVUS.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- ceVUS With the Use of OPTISON & VCUG in the Same Session: OPTISON will be resuspended just before the performance of ceVUS examination, and 0.1%-0.5% OPTISON solution will be used for intravesical administration. The exact OPTISON dose (ml) will be adjusted according to the age-related bladder filling capacity with het maximum dose (ml) range from 0.3 mL in newborns to 3 mL in 18 year-old children. VCUG exam as part of the standard care will be performed using the same bladder catheter with intravesical administration of the x-ray contrast agent.
Arm/Group | ceVUS With the Use of OPTISON & VCUG in the Same Session
Number analyzed (Participants) | 30
percentage
  sensitivity | 91.7 [61.5 to 99.8]
  specificity | 98.0 [89.4 to 99.9]
  positive predictive value | 91.7 [61.1 to 98.7]
  negative predictive value | 98.0 [88.2 to 99.7]

ADVERSE EVENTS:
Time Frame: During 48 hours following the study participation
Arm/Group | ceVUS With the Use of OPTISON & VCUG in the Same Session
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ceVUS With the Use of OPTISON & VCUG in the Same Session (N=30)
Dysuria (Renal and urinary disorders) | 1 (1) — The dysuria was an anticipated adverse event and it was categorized as mild in severity, subacute in onset and self-limited in course. No medical consultation, no medication or other intervention was required or performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes